CLINICAL TRIAL: NCT03888742
Title: A Cross Sectional Study to Assess the Effect of Androgen Deprivation Therapy on Gut and Urinary Microbiota in Patients With Prostate Cancer
Brief Title: The Effect of Androgen Deprivation Therapy on Gut and Urinary Microbiota in Patients With Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chi Fai NG, Professor, Chinese University of Hong Kong
Other Study IDs: CRE 2018.280
Record Dates: First submitted 2019-03-21; First posted 2019-03-25 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Total bacterial DNA was extracted from fecal / urine samples by using the bead-beating method with Qiagen QIAamp DNA Microbiome kit. Extracted DNA will be quantified by Nanodrop for PCR reaction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ADT Group: Participants received continue ADT treatment for at least more than 6 months
- RRP Group: Participants have radical prostatectomy performed more than 6 months ago.

SUMMARY:
The incidence of prostate cancer is increasing in Hong Kong, as well as that of recurrent or metastatic prostate cancer. Androgen deprivation therapy (ADT) is the standard treatment for recurrent or metastatic prostate cancer, with side effects such as obesity, type 2 diabetes mellitus, metabolic syndrome, osteoporosis and cognitive impairment. With the improvement of treatment, the 5-year survival rate of recurrent and metastatic prostate cancer is up to 20%, and therefore increases the chances of developing such side effects.

Due to the introduction of next generation sequencing, investigators have more knowledge of the microbiota in our body, particularly the gut microbiota. Different studies have related gut dysbiosis with obesity, type 2 diabetes mellitus and metabolic syndrome. If investigators can show that ADT is leading to gut dysbiosis, this could be a way in preventing or treating the side effects of ADT.

This study aims to identify whether ADT in patients with prostate cancer will have different composition in their gut and urine microbiota.

DETAILED DESCRIPTION:
The prostate gland is a clinically important male accessory sex gland and vital for its production of semen. Prostate cancer (PCa) is now ranked 3th in annual incidence of male cancer and ranked 5th for cancer-related death in men in Hong Kong which accounts for about 10.9 deaths per 100,000 persons. (Hong Kong Cancer registry 2015) Its incidence is rising rapidly, almost tripled in the past 10 years. As the elderly population continues to increase, the impact of PCa on the men's health and also the burden on health care system will continue to rise.

Despite the improvement in awareness of the disease and also increasing use of serum prostate specific antigen, many patients still presented at a late stage that beyond cure by local therapy. Together with those patients suffered recurrent disease after local therapy,1 many PCa patients required the use of androgen deprivation therapy (ADT) for the control of disease.

However, unlike other malignancy, PCa is characterized by its slow progression nature and even for metastatic disease the 5-year survival is upto 20%. Therefore, while ADT can provide effective control of disease, there are increasing evidences suggesting that it can also result in many adverse effects in the patients, and these effects are particular important due to the long survival of these patients. From the western literature, the adverse effects can be quite diverse.2 Classical side effects after ADT include mood changes, hot flushes, change in cognitive function,3 loss of libido, erectile dysfunction, osteoporosis and pathological fracture.4 Also there are more and more evidences showed ADT will also altered the metabolic and cardiovascular status of the patients and resulted in increase in insulin resistance and increase in risk of cardiovascular related mortality.5-7 Similarly, from our local data, investigators also observed similar increase in adverse events also happened in Chinese patients treated with ADT.8

There are many possible mechanisms proposed for the occurrence of these adverse events in patients receiving ADT, including increase in obesity, dyslipidaemia, insulin resistance etc. All these factors will lead to increase in metabolic and cardiovascular risk. However, the exact link between of hypogonadism and the development of obesity, dyslipidaemia and insulin resistance was still unclear.

Since the development of the next-generation sequencing, the knowledge of the microbiota in different sites made much progress. Of all other sites, the gut was the most frequently studied. It was found that a number of different conditions were associated with the composition of the gut microbiota, like age9, environmental factors (e.g. diet10-12), medications and diseases like obesity13, inflammatory bowel disease14 and colorectal cancer.15 Other than those mentioned, gender difference in gut microbiota was found in animal studies16 as well as human studies.17-20

On the other hand, urinary microbiota was also found to have gender differences21. The mechanism of this difference is proposed by animal studies to be related to sex hormone16,22, and it was proposed to be due to the hormone-microbe interaction, or due to the sex-specific immune response.23

Recent studies has suggested castration will affect the guts microflora and resulted in the development of obesity in mice.22 However, whether similar effect in human was unknown. Moreover, if the microflora in men was also changed by ADT, this might be one of the underlying mechanism for the increase in cardiovascular and metabolic risk observed in men receiving ADT. Therefore, investigators would like to perform a prospective study to examine the relationship between ADT and gut and urinary microbiota, and also the possible relationship with the development of metabolic and cardiovascular complications in our local population.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with age greater than or equal to 18 years old, who are able to provide consent
* Patients who was diagnosed to have prostate cancer
* Patients either received continue ADT treatment for at least more than 6 months or have radical prostatectomy performed more than 6 months ago.

Exclusion Criteria:

* Recent use of antibiotics within one month
* History of urinary tract infection in preceding year

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300 Patients (150 patients with ADT usage and 150 patients with radical prostatectomy done) who fulfilled the above inclusion criteria with no exclusion criteria will be recruited for the study.
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
Difference in the composition of gut microbiome in prostate cancer patients with or without ADT | Baseline (one-time point only)
  Total bacterial DNA was extracted from fecal / urine samples by using the bead-beating method with Qiagen QIAamp DNA Microbiome kit. Extracted DNA will be quantified by Nanodrop for PCR reaction.
Difference in the composition of urinary microbiome in prostate cancer patients with or without ADT | Baseline (one-time point only)
  Total bacterial DNA was extracted from fecal / urine samples by using the bead-beating method with Qiagen QIAamp DNA Microbiome kit. Extracted DNA will be quantified by Nanodrop for PCR reaction.

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fai NG, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fang LC, Merrick GS, Wallner KE. Androgen deprivation therapy: a survival benefit or detriment in men with high-risk prostate cancer? Oncology (Williston Park). 2010 Aug;24(9):790-6, 798. PMID 20923031
- [Background] Taylor LG, Canfield SE, Du XL. Review of major adverse effects of androgen-deprivation therapy in men with prostate cancer. Cancer. 2009 Jun 1;115(11):2388-99. doi: 10.1002/cncr.24283. PMID 19399748
- [Background] Beauchet O. Testosterone and cognitive function: current clinical evidence of a relationship. Eur J Endocrinol. 2006 Dec;155(6):773-81. doi: 10.1530/eje.1.02306. PMID 17132744
- [Background] Lattouf JB, Saad F. Bone complications of androgen deprivation therapy: screening, prevention, and treatment. Curr Opin Urol. 2010 May;20(3):247-52. doi: 10.1097/MOU.0b013e32833835be. PMID 20224416
- [Background] Smith MR. Androgen deprivation therapy and risk for diabetes and cardiovascular disease in prostate cancer survivors. Curr Urol Rep. 2008 May;9(3):197-202. doi: 10.1007/s11934-008-0035-y. PMID 18765113
- [Background] Saylor PJ, Smith MR. Metabolic complications of androgen deprivation therapy for prostate cancer. J Urol. 2009 May;181(5):1998-2006; discussion 2007-8. doi: 10.1016/j.juro.2009.01.047. Epub 2009 Mar 14. PMID 19286225
- [Background] Teoh JY, Chiu PK, Chan SY, Poon DM, Cheung HY, Hou SS, Ng CF. Risk of new-onset diabetes after androgen deprivation therapy for prostate cancer in the Asian population. J Diabetes. 2015 Sep;7(5):672-80. doi: 10.1111/1753-0407.12226. Epub 2014 Dec 22. PMID 25266491
- [Background] Vemuri R, Gundamaraju R, Shastri MD, Shukla SD, Kalpurath K, Ball M, Tristram S, Shankar EM, Ahuja K, Eri R. Gut Microbial Changes, Interactions, and Their Implications on Human Lifecycle: An Ageing Perspective. Biomed Res Int. 2018 Feb 26;2018:4178607. doi: 10.1155/2018/4178607. eCollection 2018. PMID 29682542
- [Background] David LA, Maurice CF, Carmody RN, Gootenberg DB, Button JE, Wolfe BE, Ling AV, Devlin AS, Varma Y, Fischbach MA, Biddinger SB, Dutton RJ, Turnbaugh PJ. Diet rapidly and reproducibly alters the human gut microbiome. Nature. 2014 Jan 23;505(7484):559-63. doi: 10.1038/nature12820. Epub 2013 Dec 11. PMID 24336217
- [Background] De Filippo C, Cavalieri D, Di Paola M, Ramazzotti M, Poullet JB, Massart S, Collini S, Pieraccini G, Lionetti P. Impact of diet in shaping gut microbiota revealed by a comparative study in children from Europe and rural Africa. Proc Natl Acad Sci U S A. 2010 Aug 17;107(33):14691-6. doi: 10.1073/pnas.1005963107. Epub 2010 Aug 2. PMID 20679230
- [Background] Wu GD, Chen J, Hoffmann C, Bittinger K, Chen YY, Keilbaugh SA, Bewtra M, Knights D, Walters WA, Knight R, Sinha R, Gilroy E, Gupta K, Baldassano R, Nessel L, Li H, Bushman FD, Lewis JD. Linking long-term dietary patterns with gut microbial enterotypes. Science. 2011 Oct 7;334(6052):105-8. doi: 10.1126/science.1208344. Epub 2011 Sep 1. PMID 21885731
- [Background] Gomes AC, Hoffmann C, Mota JF. The human gut microbiota: Metabolism and perspective in obesity. Gut Microbes. 2018 Jul 4;9(4):308-325. doi: 10.1080/19490976.2018.1465157. Epub 2018 May 24. PMID 29667480
- [Background] Ni J, Wu GD, Albenberg L, Tomov VT. Gut microbiota and IBD: causation or correlation? Nat Rev Gastroenterol Hepatol. 2017 Oct;14(10):573-584. doi: 10.1038/nrgastro.2017.88. Epub 2017 Jul 19. PMID 28743984
- [Background] Tilg H, Adolph TE, Gerner RR, Moschen AR. The Intestinal Microbiota in Colorectal Cancer. Cancer Cell. 2018 Jun 11;33(6):954-964. doi: 10.1016/j.ccell.2018.03.004. Epub 2018 Apr 12. PMID 29657127
- [Background] Mueller S, Saunier K, Hanisch C, Norin E, Alm L, Midtvedt T, Cresci A, Silvi S, Orpianesi C, Verdenelli MC, Clavel T, Koebnick C, Zunft HJ, Dore J, Blaut M. Differences in fecal microbiota in different European study populations in relation to age, gender, and country: a cross-sectional study. Appl Environ Microbiol. 2006 Feb;72(2):1027-33. doi: 10.1128/AEM.72.2.1027-1033.2006. PMID 16461645
- [Background] Org E, Mehrabian M, Parks BW, Shipkova P, Liu X, Drake TA, Lusis AJ. Sex differences and hormonal effects on gut microbiota composition in mice. Gut Microbes. 2016 Jul 3;7(4):313-322. doi: 10.1080/19490976.2016.1203502. Epub 2016 Jun 29. PMID 27355107
- [Background] Haro C, Rangel-Zuniga OA, Alcala-Diaz JF, Gomez-Delgado F, Perez-Martinez P, Delgado-Lista J, Quintana-Navarro GM, Landa BB, Navas-Cortes JA, Tena-Sempere M, Clemente JC, Lopez-Miranda J, Perez-Jimenez F, Camargo A. Intestinal Microbiota Is Influenced by Gender and Body Mass Index. PLoS One. 2016 May 26;11(5):e0154090. doi: 10.1371/journal.pone.0154090. eCollection 2016. PMID 27228093
- [Background] Yurkovetskiy L, Burrows M, Khan AA, Graham L, Volchkov P, Becker L, Antonopoulos D, Umesaki Y, Chervonsky AV. Gender bias in autoimmunity is influenced by microbiota. Immunity. 2013 Aug 22;39(2):400-12. doi: 10.1016/j.immuni.2013.08.013. PMID 23973225
- [Background] Markle JG, Frank DN, Mortin-Toth S, Robertson CE, Feazel LM, Rolle-Kampczyk U, von Bergen M, McCoy KD, Macpherson AJ, Danska JS. Sex differences in the gut microbiome drive hormone-dependent regulation of autoimmunity. Science. 2013 Mar 1;339(6123):1084-8. doi: 10.1126/science.1233521. Epub 2013 Jan 17. PMID 23328391
- [Background] Fouts DE, Pieper R, Szpakowski S, Pohl H, Knoblach S, Suh MJ, Huang ST, Ljungberg I, Sprague BM, Lucas SK, Torralba M, Nelson KE, Groah SL. Integrated next-generation sequencing of 16S rDNA and metaproteomics differentiate the healthy urine microbiome from asymptomatic bacteriuria in neuropathic bladder associated with spinal cord injury. J Transl Med. 2012 Aug 28;10:174. doi: 10.1186/1479-5876-10-174. PMID 22929533
- [Background] Harada N, Hanaoka R, Hanada K, Izawa T, Inui H, Yamaji R. Hypogonadism alters cecal and fecal microbiota in male mice. Gut Microbes. 2016 Nov;7(6):533-539. doi: 10.1080/19490976.2016.1239680. Epub 2016 Sep 22. PMID 27656762
- [Background] Tetel MJ, de Vries GJ, Melcangi RC, Panzica G, O'Mahony SM. Steroids, stress and the gut microbiome-brain axis. J Neuroendocrinol. 2018 Feb;30(2):10.1111/jne.12548. doi: 10.1111/jne.12548. PMID 29024170